CLINICAL TRIAL: NCT03886896
Title: Efficacy of Intravenous Lidocaine Infusion on Pain Relief in Children Undergoing Laparoscopic Appendectomy: Randomized Controlled Trial.
Brief Title: Intravenous Lidocaine in Children Undergoing Laparoscopic Appendectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Maciej Kaszyński, Principal Investigator, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Lido01
Record Dates: First submitted 2019-03-15; First posted 2019-03-22 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Acute Appendicitis; Postoperative Pain; Postoperative Nausea and Vomiting
Keywords: systemic lidocaine; nalbuphine; postoperative pain; multimodal analgesia; laparoscopic appendectomy; laparoscopy; recovery
MeSH Terms: conditions — Appendicitis; Pain, Postoperative; Postoperative Nausea and Vomiting | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A - lidocaine group (Experimental): Group A: children receiving standard general anesthesia with intravenous lidocaine infusion 1,5 mg/kg for 5 minutes before induction of anesthesia. After 5 minutes, lidocaine infusion continued at rate of 1.5 mg/kg/h during operation, and discontinued before move the patients to PACU.
  Interventions: Drug: Lidocaine
- Group B - control group (No Intervention): Group B: children receiving standard general anesthesia (involving fentanyl and sevoflurane) without lidocaine infusion

INTERVENTIONS:
Drug: Lidocaine — Lidocaine infusion during surgery
  Other Names: Intravenous lidocaine infusion
  Arms: Group A - lidocaine group

SUMMARY:
Intravenous lidocaine - a potent local anesthetic with analgesic and anti-inflammatory properties has been shown to be an effective adjunct that reduces intra and postoperative opioid consumption and facilitates pain management in adults. In children population promising but limited evidence is available. The study was planned to evaluate the efficacy of continuous intravenous infusion of lidocaine to reduce opioid consumption during and after laparoscopic appendectomy in children.

DETAILED DESCRIPTION:
Postoperative pain in children is still one of the most under diagnosed and under treated medical problems. It affects post-surgery recovery, mortality and morbidity, limits mobility. Untreated pain not only causes child's suffering but can decrease the pain threshold in the future or lead to the development of chronic pain. Postoperative analgesia has been traditionally based on opioids but as their use can be associated with adverse effects prolonging hospital stay and affecting recovery current guidelines focus on multimodal approaches involving numerous analgesics with different mechanism of action. Growing evidence suggests that intravenous lidocaine reduces intra- and postoperative requirement for opioids. Lidocaine has been proved to have analgesic and anti-inflammatory properties. It is also a potent peripheral nervous system modulator inhibiting peripheral and central sensitization. The studies performed in adult population have proved the efficacy of systemic lidocaine in postoperative pain treatment. It is an effective adjunct that reduces opioids consumption and facilitates pain management. As such lidocaine infusion has been included in postoperative pain management guidelines for adults. Studies on children population have promising results but high quality randomized controlled trials are still missing.

The proposed study has been planned to evaluate the efficacy of continuous infusion of lidocaine as an adjunct to standard general anesthesia (involving fentanyl and sevoflurane) in reducing opioids consumption and facilitating postoperative pain control in children undergoing laparoscopic appendectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 months and 18 year-old
2. Patients with American Society of Anaesthesiologists physical status (ASA) class 1/1E, 2/2E, 3/3E
3. Patients undergoing laparoscopic appendectomy

Exclusion Criteria:

1. Allergy to local anesthetics or contraindication to use of lidocaine
2. Patients with American Society of Anaesthesiologists physical status (ASA) IV or more.
3. Severe cardiovascular disease
4. Preoperative bradycardia
5. Preoperative atrioventricular block
6. Renal failure
7. Chronic treatment with analgesics
8. Parents' refusal

Ages: 18 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 74 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-17 (Actual)

PRIMARY OUTCOMES:
Postoperative opioid consumption | 24 hours after surgery
  Total nalbuphine requirement in milligrams during the first 24 hours after surgery

SECONDARY OUTCOMES:
Intraoperative opioid consumption | Intraoperative - from induction of anesthesia to extubation
  Intraoperative fentanyl consumption - amount of fentanyl in micrograms/kilogram participant's body weight
Intraoperative volatile anesthetic consumption | Intraoperative - from induction of anesthesia to extubation
  Intraoperative sevoflurane consumption in milliliters. Investigators use a standard protocol of fresh gas flow.
Time to first perception of significant pain | 24 hours after surgery
  Time to first dose of nalbuphine - pain score > 3 points. Assessing Face - Legs - Activity - Crying - Consolability Scale/Numerical Rating Scale/Visual Analog Pain Scale depending on participant's age.
Incidence of postoperative nausea and vomiting (PONV) | 24 hours after surgery
  Evaluated on a four-point ordinal scale. 0 = none, 1 = nausea, 2 = vomiting 1/hr, 3 = vomiting > 1/hr
Side effects of lidocaine will be documented | 24 hours after surgery
  Number of Participants with: headedness, tinnitus, perioral numbness, arrythmia.

CONTACTS AND LOCATIONS:
Overall Officials: Maciej Kaszyński, Principal Investigator — Medical University of Warsaw
Locations (1):
- University Clinic Centre of Medical University of Warsaw, Warsaw, Poland

REFERENCES:
- [Derived] Kaszynski M, Stankiewicz B, Palko KJ, Darowski M, Pagowska-Klimek I. Impact of lidocaine on hemodynamic and respiratory parameters during laparoscopic appendectomy in children. Sci Rep. 2022 Aug 18;12(1):14038. doi: 10.1038/s41598-022-18243-3. PMID 35982198
- [Derived] Kaszynski M, Lewandowska D, Sawicki P, Wojcieszak P, Pagowska-Klimek I. Efficacy of intravenous lidocaine infusions for pain relief in children undergoing laparoscopic appendectomy: a randomized controlled trial. BMC Anesthesiol. 2021 Jan 5;21(1):2. doi: 10.1186/s12871-020-01218-0. PMID 33397287